CLINICAL TRIAL: NCT01658995
Title: Management of Etonogestrel Subdermal Implant-related Bleeding in US Women: a Prospective, Randomized, Placebo-controlled Trial.
Brief Title: Management of Etonogestrel Subdermal Implant-related Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Petra M. Casey (Other)
Responsible Party: Sponsor-Investigator, Petra M. Casey, Associate Professor of Obstetrics - Gynecology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-008933
Record Dates: First submitted 2012-08-02; First posted 2012-08-07 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: ESI-related Bleeding
Keywords: Implanon; Etonogestrel subdermal implant; Nexplanon; Contraception; Irregular Bleeding; Menometrorrhagia
MeSH Terms: interventions — Doxycycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Post ESI implant - Doxycycline (Active Comparator): Subjects will be randomized into this arm after experiencing dissatisfaction with bleeding after 13 weeks post ESI insertion and received Doxycycline 100 mg oral capsules, twice daily for 10 days. After 10 days, subsequent treatment can requested by the subjects
  Interventions: Drug: Doxycycline
- Post ESI implant - Placebo (Placebo Comparator): Subjects will be randomized into this arm after experiencing dissatisfaction with bleeding after 13 weeks post ESI insertion and received placebo 100 mg oral capsules, twice daily for 10 days. After 10 days, subsequent treatment can requested by the subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 100 mg oral capsules twice daily for 10 days. After 10 days, an additional Secondary treatment may be requested.
  Other Names: Adoxa, Alodox, Avidoxy, Bio-Tab, Doryx, Doxy Lemmon, Doxy-Caps, Monodox, Morgidox, Ocudox, Oracea, Oraxyl, Periostat, Vibra-Tabs, Vibramycin
  Arms: Post ESI implant - Doxycycline
Drug: Placebo — Placebo, one capsule orally twice daily for 10 days. After 10 days, an additional Secondary treatment may be requested.
  Other Names: Sugar pill
  Arms: Post ESI implant - Placebo

SUMMARY:
This is a double-blinded, randomized, prospective placebo-controlled clinical trial to be conducted within the Mayo Clinic and the Mayo Clinic Health System.

The goal of the research study is to gather information to determine whether Doxycycline is effective for the treatment of unacceptable bleeding associated with the etonogestrel subdermal implant (ESI), as compared to placebo.

DETAILED DESCRIPTION:
ESI is a long-acting reversible contraceptive. Though safety and efficacy have been established world wide, only about 1 % of women have been reported to use this method. Its use is limited by bleeding pattern changes which result in requests for early removal, most commonly within the first 8 months of use.

Women ages 18-51 years, choosing ESI and who meet eligibility criteria, will be offered enrollment in the study at the time of ESI insertion. Every effort will be made to insert Implanon on the same day as consent unless medically contraindicated. Prospective diaries will be completed starting on the date of ESI insertion. All participants will be contacted by study personnel 13 weeks after enrollment and queried as to the presence of unacceptable bleeding. Bleeding concerns will be objectively assessed using a modification of the Pictorial Blood Loss Assessment Chart (PBLAC).

Participants initiating contact with bleeding concerns at any time after 13 weeks post-ESI insertion will be offered treatment randomization at the time of contact. The basis for randomized treatment will be whether the bleeding is considered "unacceptable" to the participant. This is inherently subjective, but constitutes the basis for most removal requests. Participants that report unacceptable bleeding at 13 weeks post-ESI insertion, and those who call with bleeding concerns anytime after 13 weeks post-ESI insertion, will be randomized into one of two groups, Doxycycline or matching placebo.

Participants that do not report unacceptable bleeding will continue to complete diaries and may be eligible for randomized treatment if unacceptable bleeding develops.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, aged 18-51 years
* Expressed desire for compliance-independent contraception
* No current pregnancy or anticipated desire for childbearing within 3 years of study enrollment and Implanon insertion
* Agreement to participate in all study related procedures and evaluations as documented by a signed informed consent

Exclusion Criteria:

* Current or prior use of Implanon
* Current long-term use of Doxycycline for other indications
* Known structural uterine abnormalities such as polyp, submucosal leiomyoma
* Prior permanent sterilization or endometrial ablation
* Pregnancy or desire for childbearing within 3 years
* Contraindications to or intolerance of etonogestrel
* Allergy to or intolerance of Doxycycline
* Inability or unwillingness to complete study related procedures and evaluations

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petra Casey, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Post ESI Implant - Doxycycline: Subjects who were randomization into this arm after experiencing dissatisfaction with bleeding after 13 weeks post ESI insertion and received Doxycycline 100 mg oral capsules, twice daily for 10 days. After 10 days subsequent treatment can requested by the subjects
- Post ESI Implant - Placebo: Subjects who were randomization into this arm after experiencing dissatisfaction with bleeding after 13 weeks post ESI insertion and received placebo 100 mg oral capsules, twice daily for 10 days. After 10 days subsequent treatment can requested by the subjects
Period: Overall Study
Arm/Group | Post ESI Implant - Doxycycline | Post ESI Implant - Placebo
Started | 42 | 40
Completed | 42 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post ESI Implant - Doxycycline | Post ESI Implant - Placebo | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (4.7) | 26.0 (6.9) | 25.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 38 | 37 | 75
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 39 | 39 | 78
  Black or African American | 2 | 0 | 2
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Secondary Treatment
Description: The proportion of subjects who requested additional secondary treatment of intervention after ESI
Time Frame: After initial treatment up to 39 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Post ESI Implant - Doxycycline | Post ESI Implant - Placebo
Number analyzed (Participants) | 42 | 40
Participants | 20 | 23
Statistical Analysis 1: Comparison: Post ESI Implant - Doxycycline vs Post ESI Implant - Placebo; Test type: Superiority; p = 0.37, Chi-squared; Risk Difference (RD) = -9.9, 95% CI 2-sided [-31.4 to 11.6]

2. Secondary Outcome: Subject Satisfaction
Description: Number of subjects who reported satisfaction with bleeding after 13 weeks post ESI insertion. As measured by the number of subjects answering very satisfied or satisfied on the Patient Satisfaction Survey question "To what extent have you been satisfied overall while using the contraceptive implant? Very satisfied, satisfied, neither satisfied or dissatisfied, dissatisfied or very dissatisfied."
Time Frame: 13 weeks post-treatment
Population: In Doxycycline arm 8 subjects were lost to follow up and did not complete any surveys after randomized to treatment. In Placebo arm 7 subjects were lost to follow up and did not complete any surveys after randomized to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Post ESI Implant - Doxycycline | Post ESI Implant - Placebo
Number analyzed (Participants) | 34 | 33
Participants | 15 | 17
Statistical Analysis 1: Comparison: Post ESI Implant - Doxycycline vs Post ESI Implant - Placebo; Test type: Superiority; p = 0.46, Chi-squared

3. Secondary Outcome: Removal of ESI
Description: Number of subjects who requested ESI removal
Time Frame: 26 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Post ESI Implant - Doxycycline | Post ESI Implant - Placebo
Number analyzed (Participants) | 42 | 40
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline (ESI implant) to end of study, approximately 39 weeks.
Arm/Group | Post ESI Implant - Doxycycline | Post ESI Implant - Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT01658995/Prot_SAP_000.pdf